CLINICAL TRIAL: NCT05929781
Title: Turning Pattern of Different Body Segments During Turns and Turning Performance in Healthy Adults and People With Parkinson's Disease
Brief Title: Turning Pattern of Different Body Segments During Turns and Turning Performance
Status: Completed | Type: Observational
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Other Study IDs: NYCU112100AE
Record Dates: First submitted 2023-06-21; First posted 2023-07-03 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Turning; Inter-segmental coordination; En bloc turning; Turning performance
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Young healthy adults: 1. 20-39 years old
- Middle to older healthy adults: 1. 40-80 years old
  2. age-matched with People with Parkinson's disease group
- People with Parkinson's disease: 1. 40-80 years old
  2. Diagnosis of idiopathic Parkinson's disease
  3. Hoehn and Yahr stage 1-2

SUMMARY:
This is a cross-sectional exploratory study. A total of 25 people with PD, 25 young healthy adults, and 25 middle to older adults will be recruited. Axial segment turning pattern and turning performance will be evaluated in two visits using the Vicon 3D motion analysis system, Gaitup, and 3D motion camera. The independent variables are the initiation timing of the head, upper trunk, pelvis, ankle, and foot when turning and the initiation sequence of turning (% turn). The dependent variables are turning performance, including turning velocity, turning steps, turning step length, turning step width), and stance phase (%).

DETAILED DESCRIPTION:
The first aim of the present study is to explore the correlation between axial segment turning pattern and turning performance in people with PD and healthy adults.

The second aim is to verify the validity and reliability of 3D motion camera in turning evaluation.

A total of 25 people with PD, 25 young healthy adults, and 25 middle to older adults will be recruited.

Axial segment turning pattern and turning performance will be evaluated in two visits using the Vicon 3D motion analysis system, Gaitup, and 3D motion camera.

The independent variables are the initiation timing of the head, upper trunk, pelvis, ankle, and foot when turning and the initiation sequence of turning (% turn). The dependent variables are turning performance, including turning velocity, turning steps, turning step length, turning step width), and stance phase (%).

For the data analysis, the Shapiro-Wilk test will be used to check for normal distribution. Pearson's correlation coefficient or Spearman's rank correlation coefficient will be used to examine the correlations between axial segment initiation timing and turning performance. To verify the validity and reliability, Pearson's correlation coefficient will be used for concurrent criterion validity. Intraclass correlation one-way random model will be used for test-retest reliability, showed with intraclass correlation coefficient and 95% confidence interval. A p-value of less than 0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Able to walk 5 meters without assistance device
* Able to turn independently

Exclusion Criteria:

* With neurological disorders
* MMSE< 24
* Any systemic and musculoskeletal disturbances or other causes of walking inability

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Young healthy adults
  2. Middle to older adults
  3. People with Parkinson's disease
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-07-21 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Initiation timing (sec) | Change from baseline at one week
  Initiation timing of the head, upper trunk, pelvis, ankle, and foot when turning
Turning velocity (cm/sec) | Change from baseline at one week
Turning steps | Change from baseline at one week
Turning step length (cm) | Change from baseline at one week
Turning step width (cm) | Change from baseline at one week
Stance phase (%) | Change from baseline at one week

CONTACTS AND LOCATIONS:
Overall Officials: Yea-Ru Yang, Ph.D., Study Chair — Department of Physical Therapy and Assistive Technology, National Yang Ming Chiao Tung University
Locations (1):
- Department of Physical Therapy and Assistive Technology, National Yang Ming Chiao Tung University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
This is a preliminary study and also with small sample size, so currently no plan to share data with other researchers